CLINICAL TRIAL: NCT03992755
Title: A Global, Open-Label Extension Study for Participants in LIQ861 Trials to Evaluate the Long-term Safety of Inhaled LIQ861 (Treprostinil) in Pulmonary Arterial Hypertension (WHO Group 1) Patients
Brief Title: Extension Study for Participants in LIQ861 Trials to Evaluate the Long-term Safety of Dry Powder Inhalation of Treprostinil
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Liquidia Technologies, Inc. (Industry)
Collaborators: Nuventra, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LTI-302
Record Dates: First submitted 2019-06-05; First posted 2019-06-20 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Primary Pulmonary Hypertension
Keywords: Pulmonary Arterial Hypertension; Idiopathic Pulmonary Arterial Hypertension; Heritable Pulmonary Arterial Hypertension; Drug Induced Pulmonary Arterial Hypertension; Toxin Induced Pulmonary Arterial Hypertension; Connective tissue disease
MeSH Terms: conditions — Familial Primary Pulmonary Hypertension; Pulmonary Arterial Hypertension; Connective Tissue Diseases

STUDY DESIGN:
Intervention Model Description: The study will evaluate the long-term safety of LIQ861 in PAH (WHO Group 1) patients who have completed a Liquidia LIQ861 clinical study. All patients will be treated on an outpatient basis until regulatory approval of LIQ861 or study is terminated by sponsor. Study enrollment will occur after final assessments from a prior study have been completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- LIQ861 Inhaled Treprostinil (Experimental): LIQ861 inhaled treprostinil at capsule strengths of 25 μg, 50 μg, 75 μg and 100 μg. LIQ861 will be administered using the RS00 Model 8 dry powder inhalation (DPI) device (Plastiape S.p.A.; Osnago, Italy) at dose levels of 25 μg capsule strength to 200 μg capsule strength treprostinil four times a day (QID) in individual patients. Titrating to dose levels beyond 200 μg capsule strength QID, under clinical investigator supervision, requires review and approval from the Medical Monitor.
  Interventions: Drug: LIQ861 Inhaled Treprostinil

INTERVENTIONS:
Drug: LIQ861 Inhaled Treprostinil — LIQ861 bulk powder is generated from a treprostinil/excipient matrix from which particles of precise size and shape are created and filled into a hydroxypropyl methylcellulose (HPMC) capsule (size 3). LIQ861 capsules are provided in capsule strengths of 25 μg, 50 μg, 75 μg and 100 μg treprostinil.
  Other Names: Inhaled treprostinil; Inhaled prostacyclin

SUMMARY:
The primary objective of this study is to evaluate the long-term safety of LIQ861 in patients with pulmonary arterial hypertension (PAH).

DETAILED DESCRIPTION:
One of the greatest impediments to patient treatment satisfaction with current inhaled treprostinil therapy is inconvenience. Currently, PAH patients using inhaled treprostinil may require more than 36 breaths per day using a nebulizer requiring daily set up and cleaning. The use of a discrete, hand-held dry powder inhaler to deliver treprostinil to the lungs could represent a major improvement in convenience and patient satisfaction, thereby improving the quality of life for PAH patients. Liquidia is pursuing approval of LIQ861, an inhalation dry powder formulation of treprostinil that is produced using Liquidia's PRINT® Technology (Particle Replication in Nonwetting Templates), as an alternative to current inhaled treprostinil therapy for the treatment of patients with PAH (WHO Group 1).

ELIGIBILITY:
Inclusion Criteria:

1. Evidence of a personally signed and dated informed consent document exists indicating that the patient has been informed of all pertinent aspects of the study prior to initiation of any study-related procedures.
2. Patient is willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
3. Patient has fulfilled all entry criteria at the time of enrollment in original study with LIQ861.
4. Patient has completed the protocol defined end of study procedures or met a protocol-defined and adjudicated endpoint in the original LIQ861 study in which they were enrolled.
5. Patient, whether male or female, agrees to use a medically acceptable method of contraception throughout the entire study period from informed consent through the termination visit, if the possibility of conception exists. Eligible male and female patients must also agree not to participate in a conception process (e.g., actively attempt to become pregnant or to impregnate, sperm donation, in vitro fertilization) during the study and for 30 days after the last dose of LIQ861.

Exclusion Criteria:

1. Patient prematurely discontinued LIQ861 due to a drug-related AE/SAE or tolerability issue in the original LIQ861 study in which they were enrolled, or patient did not complete protocol defined study procedures at an end of study visit (not Early Termination visit) in their original LIQ861 study.
2. Patient withdrew consent during participation in another LIQ861 study.
3. Patient is a female who wishes to become pregnant or who has a positive pregnancy test on Day 1 (LTI-302 Study Initiation Visit).
4. Patient has undergone lung or heart/lung transplant or the initiation of parenteral (intravenous [IV] infusion or subcutaneous injection) therapy with a prostacyclin during the time since participation in their original LIQ861 study.
5. Any reason exists that, in the opinion of the Investigator or Medical Monitor, precludes the patient from participating in the study, e.g., any previous or intercurrent medical condition that may increase the risk associated with study participation or that would confound study analysis or impair study participation or cooperation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2019-07-18 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment emergent adverse events (AEs). | Baseline until the end of study, approximately 2.5 years (Dec-2021).
  Treatment-emergent adverse events and serious adverse events will be grouped by MedDRA System Organ Class, dose level at onset, time on drug at onset, and relationship to dose titration.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas S Hill, MD, Principal Investigator — Tufts Medical Center
Locations (25):
- United States (25):
  - Banner University Medical Center, Phoenix, Arizona
  - Arizona Pulmonary Specialists, Ltd., Phoenix, Arizona
  - West Los Angeles VA Healthcare Center, Los Angeles, California
  - UC Davis Medical Center, Sacramento, California
  - Los Angeles Biomedical Research Center, Torrance, California
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - University of Florida, Gainesville, Florida
  - Mayo Clinic-Jacksonville, Jacksonville, Florida
  - AdventHealth, Orlando, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Northwestern Medicine, Feinberg School of Medicine, Chicago, Illinois
  - University of Chicago Medicine, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Ochsner Medical Center, New Orleans, Louisiana
  - Tufts Medical Center, Boston, Massachusetts
  - Mayo Clinic-Rochester, Rochester, Minnesota
  - University of New Mexico Health Science Center, Albuquerque, New Mexico
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Oregon Health and Science Center, Portland, Oregon
  - Alleghany General Hospital, Pittsburgh, Pennsylvania
  - UPMC Presbyterian Hospital, Pittsburgh, Pennsylvania
  - UT Southwestern Medical Center, Dallas, Texas
  - Houston Methodist Lung Center, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - INOVA Fairfax Medical Campus, Falls Church, Virginia

IPD SHARING:
Plan to Share IPD: No